CLINICAL TRIAL: NCT07202208
Title: Effectiveness of the Delirium Zero Protocol to Prevent the Onset of Delirium in Patients Undergoing Hip Fracture Surgery: Randomized Clinical Trial
Brief Title: Effectiveness of the Delirium Zero Protocol to Prevent the Onset of Delirium in Patients Undergoing Hip Fracture Surgery
Acronym: DZ
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cardenal Herrera University (Other)
Collaborators: Hospital Politècnic i Universitari la Fe de València (Unknown)
Responsible Party: Principal Investigator, Laura García Garcés, Assistant Professor, Cardenal Herrera University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: DZ_Delirum Zero; PINV_05CNDE24 (Other Grant/Funding Number: Conferencia Nacional de Decanos de Enfemería (CNDE))
Record Dates: First submitted 2025-07-22; First posted 2025-10-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Hip Fracture; Delirium - Postoperative
Keywords: hip fracture; Family; Care; Care Protocol; Delirium; Caregiver
MeSH Terms: conditions — Hip Fractures; Emergence Delirium; Delirium

STUDY DESIGN:
Intervention Model Description: Randomized Clinical Trial, simple blind, parallel, two-arm.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Delirium Zero (Experimental): In addition to the standard of care that the Control Group receives, the Intervention Group (Delirium Zero) will be subjected to the 'Delirium Zero' protocol.
  Interventions: Procedure: "Delirium Zero" protocol; Procedure: Standard of Care to prevent Delirium.
- Control Group (Active Comparator): The Control Group receives the standard of care to prevent delirium.
  Interventions: Procedure: Standard of Care to prevent Delirium.

INTERVENTIONS:
Procedure: "Delirium Zero" protocol — The protocol consists of: i) a patient orientation poster placed in the room in a visible location for the patient, with information updated daily by the family member/caregiver; ii) a clock hung on the wall next to the orientation poster; and iii) a verification sheet of the preventive measures taken by the caregiver/family member, where the caregiver/family member must indicate daily the frequency with which preventive activities have been performed. The caregiver/family member will have this document in the patient's room all day and will need to complete it at the end of the day, when the nurse will collect it for safekeeping. From that day until the patient is discharged, the nurse responsible for the patient's care will be responsible for providing a new verification sheet of the preventive measures taken by the family member/caregiver and collecting it at the end of the day once it has been completed by the family member/caregiver.
  Arms: Delirium Zero
Procedure: Standard of Care to prevent Delirium. — All participants in the study, regardless of the assigned group, receive information on strategies to prevent delirium, which is provided in the participant information sheet and includes an infographic and a guide for patients and their families. Participants are advised to keep this document accessible throughout their stay for reference.

SUMMARY:
The main objective of this research will be to investigate whether the control of care provided by the family/caregiver can prevent the onset of delirium in individuals undergoing surgical intervention for hip fracture.

The research will be a randomized, single-blind, parallel, two-arm clinical trial that compares two conditions: intervention group, hereafter IG (Delirium Zero protocol based on a space-temporal orientation poster for the patient, a clock hung on the wall next to the orientation poster, and a checklist for the preventive measures taken by the caregiver/family), and control group, hereafter CG (standard of care).

The participants will be patients over 65 years old, admitted to the trauma hospitalization units of the La Fe University and Polytechnic Hospital (La Fe Health Department, Valencia, Spain), operated on for hip fracture and accompanied by a relative/caregiver.

The research will be carried out at the La Fe University and Polytechnic Hospital (La Fe Health Department, Valencia, Spain) because it is the reference hospital for the Valencian Community, and because the rooms in this center are private, which allows for no interference between the intervention under study (in GI) or the standard care (GC).

ELIGIBILITY:
Inclusion Criteria:

* The participants will be patients over 65 years old
* Admitted to the orthopedic hospitalization units of the La Fe University and Polytechnic Hospital (La Fe health department, Valencia, Spain).
* Who are undergoing surgery for hip fracture
* Accompanied by a family member/caregiver who understands Spanish and knows how to read and write it.

Exclusion Criteria:

* Have previously been diagnosed with severe cognitive impairment according to the Pfeiffer scale, which corresponds to a score of 8-10 points.
* Have previously been diagnosed with any serious mental disorder (schizophrenic disorders, schizotypal disorders, persistent delusional disorders, substance-induced delusional disorders, schizoaffective disorders, other non-organic psychotic disorders, bipolar disorder, serious depressive episode with psychotic symptoms, and severe recurrent depressive disorders). - that they have delirium at the time of admission to the trauma room.
* That they have a language barrier, deep aphasia, coma, or terminal illness.
* That they have been previously enrolled in this study.
* That before the surgery they were admitted to a different hospital unit than those participating in the study, although they may then be transferred to one of these trauma units.
* That before entering the trauma hospitalization unit, they have been in the emergency room for more than 36 hours.
* That they present brain alterations (tumors, occupying lesions).

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2025-01-15 (Actual); Primary Completion 2028-07-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Delirium: appearance | Baseline, from the patient's admission to the trauma unit until hospital discharge or assessedup to 6 weeks, whichever came first.
  It will be measured using the Confusion Assessment Method scale. It will be measured twice daily, in the morning and in the afternoon, during all days of hospitalization, in all participants, regardless of the group they belong to.
  The scale allows for the detection of acute confusional state (delirium) using an algorithm that assesses four criteria: criterion 1 (presence of an acute and fluctuating change in the patient's mental status and behavior), criterion 2 (inattention), criterion 3 (disorganized thinking), and criterion 4 (altered level of consciousness). To establish the presence of delirium, the presence of criteria 1 and 2 is mandatory, as well as any one of criteria 3 and 4. A criterion is considered present when: the questions are answered affirmatively (for criteria 1, 2, and 3) and when the level of consciousness is other than alert (for criterion 4).

SECONDARY OUTCOMES:
Delirium: severity | Baseline, from the patient's admission to the trauma unit until hospital discharge or assessedup to 6 weeks, whichever came first.
  It will be measured using the Confusion Assessment Method scale. It will be measured twice daily, in the morning and in the afternoon, during all days of hospitalization, in all participants, regardless of the group they belong
  Based on the CAM scale, numerical scores are assigned to the evaluated criteria, which allows the intensity of the delirium symptoms to be quantified, with a score that ranges from 0 to 7, where a higher score indicates greater severity. Each of the symptoms is scored as follows: criterion 1 (acute onset and fluctuating course of mental state, rated as absent = 0, or present = 1), criterion 2 (inattention, rated as absent = 0, mild = 1 or marked = 2), criterion 3 (disorganized thinking, rated as absent = 0, mild = 1 or marked = 2) and criterion 4 (altered level of consciousness, where an alert state of consciousness is considered normal = 0, and the rest of the states are considered altered with these scores: vigilant = 1, lethargic = 1, stupor = 2, coma = 2).
Delirium. Days of duration | Baseline, from the patient's admission to the trauma unit until hospital discharge or assessedup to 6 weeks, whichever came first.
  Days of delirium. Once the patient is discharged, the principal investigator will record the total number of days the patient experienced delirium during their stay. Unit of measurement: days. Method of aggregation: absolute frequency.
  It will be measured twice daily, in the morning and in the afternoon, during all days of hospitalization, in all participants, regardless of the group they belong to.
Delirium: number of episodes | Baseline, from the patient's admission to the trauma unit until hospital discharge or assessedup to 6 weeks, whichever came first.
  Number of delirium episodes during the stay. Once the patient is discharged, the principal investigator will record the total number of delirium episodes the patient experienced during their stay. Unit of measurement: number of episodes. Method of aggregation: absolute frequency.
  It will be measured twice daily, in the morning and in the afternoon, during all days of hospitalization, in all participants, regardless of the group they belong to.
Adherence to the Delirium Zero protocol | Baseline, from the patient's admission to the trauma unit until hospital discharge or assessedup to 6 weeks, whichever came first.
  The Delirium Zero protocol is applied only to participants in the IG. Adherence to this protocol is measured by recording the frequency of delirium prevention measures.
  For each preventive measure, the frequency with which it was performed is indicated using a Likert-type scale with four frequency options: Never = 0, Sometimes = 1, Quite a bit = 2, and Always = 3. The measure of being accompanied at night by a family member/caregiver, and the measures related to poster completion, have two response options: No = 0 and Yes = 1. The score ranges from 0 to 36 in patients without glasses, hearing aids, or dentures, with higher scores indicating greater adherence to the protocol. This maximum score will be increased by 6 points for patients with glasses and/or 6 points for patients with hearing aids and/or 3 points for patients with dentures. In addition, an analysis of overall adherence will be performed.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario y Politécnico La Fe, Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No